CLINICAL TRIAL: NCT03380117
Title: Electronic Bridge to Mental Health for College Students (eBridge)
Brief Title: Electronic Bridge to Mental Health for College Students
Acronym: eBridge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Cheryl A. King, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01MH103244 (NIH)
Record Dates: First submitted 2017-11-15; First posted 2017-12-20 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Suicide; Depression
Keywords: Suicidal Ideation; Suicide Attempt; Risk Screening; Online Intervention; Online Counseling; College Students; Motivational Interviewing; Linkage to Care
MeSH Terms: conditions — Suicide; Depression; Suicidal Ideation; Suicide, Attempted

STUDY DESIGN:
Intervention Model Description: In eBridge, students take an online screen and receive personalized feedback about their self-reported depression, alcohol/substance use, and level of functioning. Students are randomly assigned to either the eBridge or control condition. In the eBridge condition, personalized feedback is provided in a graphic format that is accompanied by motivational-interviewing-adherent statements. In this condition, students' communications with eBridge counselors will occur via online dialogues, in which students and counselors exchange messages using a secure website. In the control condition, personalized feedback will also be delivered online to students, highlighting their personal data and specify links between key screening variables and negative outcomes. However, in the control condition, this is provided in a straightforward graphic, informational format, which is consistent with standard practice in online screening programs for college students.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eBridge Online Counseling (Experimental): In the eBridge condition, personalized feedback is provided in a graphic format that is accompanied by motivational-interviewing-adherent statements. In this condition, students have the opportunity to engage with eBridge counselors via online dialogues, in which students and counselors exchange messages using a secure website.
  Interventions: Behavioral: eBridge Online Counseling
- Control (No Intervention): In the control condition, personalized feedback will also be delivered online to students, highlighting their personal data and specify links between key screening variables and negative outcomes. However, in the control condition, this is provided in a straightforward graphic, informational format, which is consistent with standard practice in online screening programs for college students.

INTERVENTIONS:
Behavioral: eBridge Online Counseling — In eBridge, students take an online screen and receive personalized feedback about their self-reported depression, alcohol/substance use, and level of functioning. Students are randomly assigned to either the eBridge or control condition. In the eBridge condition, personalized feedback is provided in a graphic format that is accompanied by motivational-interviewing-adherent statements. In this condition, students' communications with eBridge counselors will occur via online dialogues, in which students and counselors exchange messages using a secure website. In the control condition, personalized feedback will also be delivered online to students, highlighting their personal data and specify links between key screening variables and negative outcomes. However, in the control condition, this is provided in a straightforward graphic, informational format, which is consistent with standard practice in online screening programs for college students.
  Arms: eBridge Online Counseling

SUMMARY:
Electronic Bridge to Mental Health for College Students (eBridge) is an online intervention that screens students for mental health concerns that include elevated suicide risk and facilitates their linkage to mental health (MH) services. EBridge is designed to work on computers, tablets, and smartphones (iOS, Android) and is easily adaptable to evolving technologies in the future. It incorporates motivational interviewing (MI) principles and draws from health behavior models that emphasize autonomy and self-determination. Following a web-based screen using standardized scales to identify students at elevated risk, eBridge offers students options for personalized feedback (provided online in a conversational format adherent with motivational interviewing) and corresponding online with professionals trained in motivational interviewing and knowledgeable about university and community resources. Ebridge is being conducted at four universities: the University of Michigan, the University of Nevada-Reno, the University of Iowa, and Stanford University.

DETAILED DESCRIPTION:
This randomized controlled trial will examine the efficacy of the intervention, Electronic Bridge to Mental Health for College Students (eBridge), in a large-scale, multi-university trial involving students at the University of Michigan, the University of Iowa, the University of Nevada-Reno, and Stanford University. Subject recruitment will take place in the fall academic semester during each year of data collection. All 6-month follow-up assessments will occur 5 to 6 months later and before many students leave campus for a spring or summer break. The study team will send recruitment emails between late September and October, and five to six-month follow-up emails in March or April. Student email addresses will be obtained from the registrar database of each participating university, per the standard Institutional Review Board and administrative process for obtaining such directory information for research studies. Furthermore, this process uses methods to maximize the security and confidentiality of the students' data, such as giving them unique identifiers to log into the web site (rather than identifiers that contain their name or email address) and using state-of-the-art security software to protect the website from having information intercepted. The planned number of student names and email addresses for possible participation will be randomly drawn. The study team will then send emails inviting students into the study, with up to 3 reminders spaced by 3-4 days for those who have yet to respond. The emails will note that students can reply and decline participation (and any further reminders). For those interested in participating, the email will contain a link to a secure web site where they can view the informed consent and decide whether to participate. The eBridge invitation email, screening, and all subsequent contacts via the Internet are confidential.

Personalized Feedback (PF) will be delivered online and provide feedback to students about their self-reported depression, alcohol/substance use, and level of functioning. This report is a briefer, modified version of the Personalized Feedback Report used in COMBINE, the multi-site clinical trial conducted to study the efficacy of treatments for alcohol dependence. The report highlights personal data and specifies links between our key screening variables and risk of negative outcomes. In the eBridge condition, PF is provided in a graphic format that is accompanied by MI-adherent statements. In addition, students in the eBridge condition have the option of viewing or not viewing their PF, and of choosing to observe their PF in one or more domain.

Students' communications with eBridge counselors (MI-trained mental health professionals) will occur via online dialogues, in which students and counselors exchange messages using a secure web site. The total duration of the exchanges is expected to be brief, in keeping with MI approaches used in medical settings to consider behavior change and/or treatment recommendations and as found in our R34 study. Students will be able to communicate with eBridge counselors using asynchronized communication (with email notification that response has been posted on secure website) at any time.

Personalized Feedback (PF) will also be delivered online to students in the control condition, providing information to students about their self-reported depression, alcohol/substance use, and level of functioning. As for students in the eBridge condition, it will highlight their personal data and specify links between key screening variables and negative outcomes. However, in the control condition, this is provided in a straightforward graphic, informational format, which is consistent with standard practice in online screening programs for college students (e.g., www.ulifeline.org). All students in the control condition receive their PF immediately upon completing their screening survey (automatic next screen).

Each student, regardless of study condition, will see a list of campus and community resources for mental health and alcohol/substance abuse treatment, and for crisis services. These will be presented on each webpage of both the screening survey and the PF report. The resource information list has been uploaded to this application as an additional document.

The research team will collect quantitative and qualitative data. Quantitative data will be collected from subjects using brief questionnaires at baseline, 4 weeks, and six months. A subset of questions from the baseline questionnaire will serve as the screen that determines whether subjects are eligible for randomization. The baseline questionnaire will be programmed such that, once determined that a subject does not meet criteria for randomization, he or she will not be asked any more questions. The measures will be brief, requiring approximately 2-10 minutes for completion (5-6 minutes at 4-weeks), because brevity is a determinant of response rates for Internet surveys.

Students will be assessed at 4 weeks because a subset may derive benefit from the online intervention itself. This assessment occurs following exposure to eBridge, yet before participants are likely to have started using services. This will help to ascertain whether some reduction in risk factors is due to the web-based intervention itself rather than to linkage to services. This brief assessment will consist of the three suicidal ideation/behavior items, the Patient Health Questionnaire-9 (PHQ-9), the PHQ-10 (single item), the Alcohol Use Disorders Identification Test (AUDIT), mental health service utilization items, and the readiness scale (see below). A full outcome assessment will be conducted at 6 months.

Participants will be remunerated for involvement in the study. A random drawing will take place for all who have received an invitation to participate. In addition a 4-week pre-incentive will be distributed to encourage students to participate. Finally, 4-week and 6-month incentives will be distributed upon completion of each assessment.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* currently enrolled full- or part-time at a participating university

Exclusion Criteria:

* not currently living in the university community (e.g., completing a study abroad semester)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6241 (Actual)
Dates: Start 2014-11-11 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-05-07 (Actual)

PRIMARY OUTCOMES:
Change in mental health service utilization | Baseline, 4 weeks, 6 months
  Change in the number of participants accessing mental health services include psychotherapy, psychopharmacological treatment, or a combination.
Adherence to mental health services, as measured by yes/no response for 4-week period. | 4 weeks
  Mental health services include psychotherapy, psychopharmacological treatment, or a combination.
Adherence to mental health services, as measured by total # of sessions for 4-week period. | 4 weeks
  Mental health services include psychotherapy, psychopharmacological treatment, or a combination.
Adherence to mental health services, as measured by yes/no response for 6-month period. | 6 months
  Mental health services include psychotherapy, psychopharmacological treatment, or a combination.
Adherence to mental health services, as measured by total # of sessions for 6-month period. | 6 months
  Mental health services include psychotherapy, psychopharmacological treatment, or a combination.

SECONDARY OUTCOMES:
Change in suicidal thoughts | Baseline, 4 weeks, 6 months
  Assessed using one item from the National Comorbidity Survey asking about serious suicidal thoughts at Baseline, 4-week, and 6-month intervals. "Have you ever felt so low you thought about committing suicide?" (Yes/No)
Change in suicidal thoughts | Baseline, 4 weeks, 6 months
  Assessed using one item from the National Comorbidity Survey asking about serious suicidal thoughts at Baseline, 4-week, and 6-month intervals. "Has there ever been a period of 2 weeks or more when you felt like you wanted to die?" (Yes/No).
Change in suicide attempts | Baseline, 4 weeks, 6 months
  Two items from the National Comorbidity Survey assess number of suicide attempts at Baseline, 4-week, and 6-month intervals. At Baseline, "How many times have you attempted suicide in your lifetime?" (open-text). At 4-week, and 6-month intervals, "In the past month, have you ever attempted suicide" (Yes/No)
Change in depression, as measured using the Patient Health Questionnaire (PHQ-9) | Baseline, 4 weeks, 6 months
  The PHQ-9 is a 9-item scale based on Diagnostic Statistical Manual IV criteria for a major depressive episode. The instrument asks the respondent to indicate the frequency of various symptoms over the past two weeks and, following standard interpretation algorithms, categorizes participants as screening positive for major depression or not.
Change in substance misuse | Baseline, 6 months
  Substance misuse will be assessed using five questions about recent drug use activity, using a list of commonly abused prescription drugs and illegal. The scale response options include never, once or twice, monthly, weekly, daily, or almost daily.
Change in alcohol misuse | Baseline, 4 weeks, 6 months
  Alcohol misuse will be assessed using the 10-item AUDIT, which asks about frequency of any drinking, average amount per day, and frequency of binge drinking (6 or more drinks on one occasion). It is scored on a 0-12 scale, and a screen cutoff score of 8 is considered optimal to identify students at higher risk.

OTHER OUTCOMES:
Academic performance, as measured by grade point average | 6 months
  Academic performance will be measured by grade point average at 6 months
Academic performance, as measured by retention | 6 months
  Academic performance will be measured by whether or not the participant is still enrolled in the university.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl King, Ph.D., Principal Investigator — Professor
Locations (4):
- United States (4):
  - Stanford University, Stanford, California
  - University of Iowa, Iowa City, Iowa
  - University of Michigan, Ann Arbor, Michigan
  - University of Nevada-Reno, Reno, Nevada

REFERENCES:
- [Derived] Bornheimer LA, Czyz E, Koo HJ, Li Verdugo J, Eisenberg D, Zheng K, Pistorello J, Albucher RC, Coryell W, Favorite T, King CA. Suicide risk profiles and barriers to professional help-seeking among college students with elevated risk for suicide. J Psychiatr Res. 2022 Aug;152:305-312. doi: 10.1016/j.jpsychires.2022.06.028. Epub 2022 Jun 18. PMID 35772258
- [Derived] Horwitz AG, McGuire T, Busby DR, Eisenberg D, Zheng K, Pistorello J, Albucher R, Coryell W, King CA. Sociodemographic differences in barriers to mental health care among college students at elevated suicide risk. J Affect Disord. 2020 Jun 15;271:123-130. doi: 10.1016/j.jad.2020.03.115. Epub 2020 Apr 18. PMID 32479307
- [Derived] Horwitz AG, Berona J, Busby DR, Eisenberg D, Zheng K, Pistorello J, Albucher R, Coryell W, Favorite T, Walloch JC, King CA. Variation in Suicide Risk among Subgroups of Sexual and Gender Minority College Students. Suicide Life Threat Behav. 2020 Oct;50(5):1041-1053. doi: 10.1111/sltb.12637. Epub 2020 Apr 15. PMID 32291833